CLINICAL TRIAL: NCT05299463
Title: Feasibility and Validity of Remote Exercise Testing in Patients With Pulmonary Hypertension
Brief Title: Remote Exercise Testing in Patients With Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 293065
Record Dates: First submitted 2021-06-30; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise Test

STUDY DESIGN:
Masking Description: Exercise study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other)
  Interventions: Diagnostic Test: Exercise Testing

INTERVENTIONS:
Diagnostic Test: Exercise Testing — * Tele-Six-minute walk test (T6MWT)
  * 1 Minute Sit-to-stand test (STS)
  * 2-minute symptom-limited Step test (ST)
  * 3-metre Timed up and go test (TUG).

SUMMARY:
The investigators plan to investigate the feasibility and validity of tests of exercise capacity, when these are performed in hospital and at home, by patients who are diagnosed with pulmonary hypertension.

Patients with pulmonary hypertension develop high blood pressure within the lungs, leading to a limitation in the amount of exercise they are able to perform. At diagnosis and follow-up patients routinely perform short exercise tests which are performed under supervision in the clinic or hospital. The results from these are compared over time and are used to assess how stable patients are. Currently, patients are required to travel to hospital to perform such a test and thus telephone or video appointments do not include this information. This study aims to investigate a range of exercise tests to assess whether they are valid in pulmonary hypertension (whether the results are comparable to the results from the current exercise test performed in hospital, the six-minute walk test) and whether it is feasible for patients to to perform these tests at home.

The investigators aim to investigate four different home exercise tests, including a sit-to-stand test, a timed up and go test, a six-minute walk test and a step test. The investigators will ask patients to perform these tests in a hospital environment and at home on two occasions. The results of these will be compared to see how they change over time and will be compared to other results obtained during standard care. Additionally, patients will be asked a questionnaire to assess their views on the four tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-years-old and above
* Diagnosed with pulmonary hypertension from any ERS/ESC group
* Able to give informed consent

Exclusion Criteria:

* Unable to provide consent
* Restricted so as unable to perform a standard 6MWT, either due to mobility or symptoms
* Patients feel they would be unable to perform any of the 4 study tests when at home
* Concerns about the patient's safety of performing home-based exercise tests (as decided by the consenting clinician and/or the patient)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional assessment of novel exercise test validity (part 1) | 2 years
  During the inpatient hospital visit (visit 1), correlation will be analysed between the distance (metres) walked on a six-minute walk test and the outcome of each of the study tests (as listed below).
  1. TUG - time (seconds)
  2. T6MWT - distance (metres)
  3. STS - number of steps
  4. ST - distance (metres) Correlation will be measured by Pearson's R Calculator for parametric data and Spearman's Rho for non-Parametric data.
Cross-sectional assessment of novel exercise test validity (part 2) | 2 years
  Agreement will be analysed between each of study tests when performed during visit 1 (inpatient hospital visit) and when performed during visit 2 (within 7 days of being discharged from hospital). This will be performed with Bland-Altman analysis.
Longitudinal study of feasibility | 2 years
  Proportion of patients that completed each of the allocated tests at visit 2 and at visit 3 (3 months after being discharged from hospital).
Longitudinal study of validity | 2 years
  Concordance of change will be analysed between each of study tests when performed during visit 2 (and when performed during visit 3. This degree of change will be compared against the patients standard six minute walk test result when measured at visit 1 and visit 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Scottish Pulmonary Vascular Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No